CLINICAL TRIAL: NCT00564265
Title: Outcomes of Surgical Treatment of Gastrointestinal Stromal Tumors in the IV Region of Chile
Brief Title: Current Management of Gastrointestinal Stromal Tumors (GIST) in the Region of Coquimbo
Status: Completed | Type: Observational
Sponsor: Cirujanos la Serena (Other)
Responsible Party: Sobelcru Ltda, Sobelcru Ltda
Other Study IDs: HLS-0047-11-07; 0047-11-07
Record Dates: First submitted 2007-11-26; First posted 2007-11-27 (Estimated); Results first posted 2009-10-21 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2010-09

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: GIST
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GIST: GIST from all gastrointestinal origins: esophagus, stomach, duodenum, jejunum, ileum, colon and rectum
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Not applied

SUMMARY:
This is a retrospective analysis and description of the preferred diagnostic and treatment methods employed on GIST on the Region of Coquimbo from 2003 to 2008.

ELIGIBILITY:
Inclusion Criteria:

* All operated patients with GIST
* Positive immunohistochemistry

Exclusion Criteria:

* Patients with GIST not operated
* Patients with GIST operated on but without immunohistochemistry

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients operated on for GIST
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo A Beltran, MD, Principal Investigator — Hospital de La Serena
Locations (1):
- Hospital De La Serena, La Serena, Coquimbo Region, Chile

REFERENCES:
- See also: Revista Chilena de Cirugia, 2011; 63:290-296 — http://www.scielo.cl/pdf/rchcir/v63n3/art09.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospital patients operated on for Gastrointestinal stromal tumor (GIST)
Pre-assignment Details: The intention was to include all consecutive patients with GIST who presented during the study period. All consecutive patients with GIST were included during the study period
Groups:
- Gastrointestinal Stromal Tumor (GIST): GIST in all locations: Stomach, duodenum, jejunum, ileum, and rectum. All patients were submitted to surgery and in 2 cases are on Imatinib therapy.
Period: Overall Study
Arm/Group | Gastrointestinal Stromal Tumor (GIST)
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gastrointestinal Stromal Tumor (GIST)
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 49 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Region of Enrollment [Number; unit: participants]
  Chile | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Survived
Description: The outcomes were measured through follow-up visits of the patients to the out-patient clinic of our institution at 15 days, 1 month, 3 months, 6 months, 1 year, and after that, every year after the surgical treatment.
Time Frame: 5 years
Population: This is a consecutive sample of all patients operated on for GISTs in 3 hospitals during a period of 5 years. The period of 5 years was determined by the time that we count with inmunochemistry to confirm GISTs at our institutions, and that time would be the last 5 years. The Last Observation Carried Dorward (LOCF) was made in August 2008.
Measure: Number; unit: Participants
Arm/Group | Gastrointestinal Stromal Tumor (GIST)
Number analyzed (Participants) | 24
Participants | 5

ADVERSE EVENTS:
Time Frame: No adverse events were assessed or collected (0/24)
Description: Adverse events were not assessed (threshold of 0%).
Arm/Group | Gastrointestinal Stromal Tumor (GIST)
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No